CLINICAL TRIAL: NCT01439724
Title: Phase III Trial of Low-level Laser Therapy to Prevent Induced Oral Mucositis in Head and Neck Cancer Patients Submitted to Concurrent Chemoradiation
Brief Title: Low-level Laser Therapy to Prevent Oral Mucositis in Head and Neck Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INCABrazil; Protocol 17/2007 (Registry Identifier: Protocol 17/2007)
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2013-02

CONDITIONS: Squamous Cell Carcinoma of Nasopharynx; Squamous Cell Carcinoma of Oropharynx; Squamous Cell Carcinoma of Hypopharynx
Keywords: Oral mucositis; Low Level Laser Therapy; Head and neck cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Stomatitis; Head and Neck Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients in the placebo group received the same treatment during the same time, but in this case the laser tip produced no light.
  Interventions: Device: Placebo (DMC, São Paulo, Brazil)
- Low Level Laser Therapy (Experimental): The investigators used a Low Level Laser Therapy, diode laser (DMC, São Paulo, Brazil) InGaAlP (indium phosphide, gallium and aluminum), with 100mW, 4J/cm ², with an area of 0.24 cm ². The laser was daily applied by a dentist and touched the mucosa of the lips, right and left buccal mucosa, left and right lateral tongue border, buccal floor and ventral tongue, totaling nine points per region.
  Interventions: Device: Low Level Laser Therapy- (DMC, São Paulo, Brazil)

INTERVENTIONS:
Device: Low Level Laser Therapy- (DMC, São Paulo, Brazil) — Diode laser (DMC,São Paulo, Brazil) InGaAlP (indium phosphide, gallium and aluminum), with 100 mW, 4J/cm ², with an area of 0.24 cm ². The laser was daily applied by a dentist and touched the mucosa of the lips, right and left buccal mucosa, left and right lateral tongue border, buccal floor and ventral tongue, totaling nine points per region.
  Other Names: Low Power Laser Therapy; Low Energy Laser Therapy
  Arms: Low Level Laser Therapy
Device: Placebo (DMC, São Paulo, Brazil) — The placebo (DMC, São Paulo, Brazil) was daily applied by a dentist and touched the mucosa of the lips, right and left buccal mucosa, left and right lateral tongue border, buccal floor and ventral tongue, totaling nine points per region.Patients in the placebo group received the same treatment during the same time, but in this case the laser tip produced no light.
  Other Names: Low power laser therapy; Low energy laser therapy
  Arms: Placebo

SUMMARY:
Oral mucositis remains a limiting factor in in head and neck squamous cell carcinomas patients treated with chemoradiation leading to pain, dysphagia, and weight loss. Low-level laser therapy emerges as a promising, preventive therapy of chemoradiation-induced OM. This study was designed to assess the efficacy of Low Level Laser Therapy (LLLT) in reducing the incidence and/or severity of oral mucositis.

DETAILED DESCRIPTION:
Assuming oral mucositis grade 3 for placebo 0.4 (P0); laser group 0.15 (P1) ; β=0.2; α=0.05, sample size was 94 pts. From Jun 2007 to Dec 2010, 47 laser group and 47 placebo patients bearer of head and neck squamous cell carcinomas of nasopharynx, oropharynx and hypopharynx entered a prospective, randomized, double blind, placebo-controlled, phase III trial. chemoradiotherapy consisted of conventional radiotherapy 70.2 Gray (Gy) (1.8Gy/d, 5 times/wk) + concurrent cisplatin 100 mg/m2 every 3 weeks. The primary end point was the incidence of grade 3-4 oral mucositis. The Low-level laser therapy used daily, was a diode indium phosphide, gallium and aluminum (InGaAlP), 660nm-100 milliwatts (mW)-4 Joules (J)/cm²(DMC, São Carlos, São Paulo, Brazil). Oral mucositis evaluation was done by WHO and Oral Mucositis Assessment Scale (OMAS) scale.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological diagnosis of squamous cell carcinoma (nasopharynx, oropharynx and hypopharynx)
* Candidates for surgery or treatment for organ preservation
* Performance status (PS) of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG)
* Indication for radiotherapy and concurrent platinum-based chemotherapy
* Oral mucosa intact
* Agree to follow the protocol of oral hygiene
* Informed consent.

Exclusion Criteria:

* Patients using medication for treatment and or prevention of mucositis
* Patients incapable of treatment compliance or of performing the protocol of oral hygiene

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heliton S Antunes, DDS, PhD, Principal Investigator — Instituto Nacional de Cancer, Brazil; Carlos G Ferreira, MD, PhD, Study Director — Instituto Nacional de Cancer, Brazil
Locations (1):
- Instituto Nacional de Cancer, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Antunes HS, Schluckebier LF, Herchenhorn D, Small IA, Araujo CM, Viegas CM, Rampini MP, Ferreira EM, Dias FL, Teich V, Teich N, Ferreira CG. Cost-effectiveness of low-level laser therapy (LLLT) in head and neck cancer patients receiving concurrent chemoradiation. Oral Oncol. 2016 Jan;52:85-90. doi: 10.1016/j.oraloncology.2015.10.022. Epub 2015 Nov 11. PMID 26559740

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Level Laser Therapy: The investigators used a diode laser (DMC, São Paulo, Brazil) InGaAlP (indium phosphide, gallium and aluminum), with 100mW, 4 Joules(J)/cm ², with an area of 0.24 cm ². The laser was daily applied by a dentist and touched the mucosa of the lips, right and left buccal mucosa, left and right lateral tongue border, buccal floor and ventral tongue, totaling nine points per region.
  Low Level Laser Therapy- (DMC, São Paulo, Brazil): Diode laser (DMC,São Paulo, Brazil) InGaAlP (indium phosphide, gallium and aluminum), with 100 mW, 4J/cm ², with an area of 0.24 cm ². The laser was daily applied by a dentist and touched the mucosa of the lips, right and left buccal mucosa, left and right lateral tongue border, buccal floor and ventral tongue, totaling nine points per region.
Period: Overall Study
Arm/Group | Placebo | Low Level Laser Therapy
Started | 47 | 47
Completed | 38 | 39
Not Completed | 9 | 8
Not completed — missing consultation | 9 | 8

BASELINE CHARACTERISTICS:
Population: The primary end point of the study was the incidence of grade 3-4 OM according to the WHO scale. Assuming an α = 0.05 and a β = 0.20, with the estimates of proportion being 0.40 for placebo (P0) and 0.15 for LLLT (P1) a total of 94 patients were evaluated.
Groups:
- Low Level Laser Therapy: The investigators used a diode laser (DMC, São Paulo, Brazil) InGaAlP (indium phosphide, gallium and aluminum), with 100 mW, 4J/cm ², with an area of 0.24 cm ². The laser was daily applied by a dentist and touched the mucosa of the lips, right and left buccal mucosa, left and right lateral tongue border, buccal floor and ventral tongue, totaling nine points per region.
  Low Level Laser Therapy- (DMC, São Paulo, Brazil): Diode laser (DMC,São Paulo, Brazil) InGaAlP (indium phosphide, gallium and aluminum), with 100 mW, 4J/cm ², with an area of 0.24 cm ². The laser was daily applied by a dentist and touched the mucosa of the lips, right and left buccal mucosa, left and right lateral tongue border, buccal floor and ventral tongue, totaling nine points per region.
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Level Laser Therapy | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (8.6) | 53.5 (6.9) | 54.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 40 | 42 | 82
Region of Enrollment [Number; unit: participants]
  Brazil | 47 | 47 | 94

OUTCOME MEASURES:

1. Primary Outcome: Incidence and / or Severity of Oral Mucositis
Description: The oral cavities of all patients were evaluated daily, from the first day until the last day of treatment. We used the scales of mucositis of the World Health Organization (WHO) and the Oral Mucositis Assessment Scale (OMAS) and a visual analogue scale (VAS) for pain assessment.
Time Frame: 7 weeks
Population: Data related to the primary endpoint were handled in a per protocol treatment analysis.
Measure: Number; unit: Grade 3-4 oral mucositis
Arm/Group | Placebo | Low Level Laser Therapy
Number analyzed (Participants) | 47 | 47
Grade 3-4 oral mucositis | 19 | 3
Statistical Analysis 1: Comparison: Placebo vs Low Level Laser Therapy; The primary end point of the study was the incidence of grade 3-4 oral mucositis (OM) according to the WHO scale. Assuming an α =0.05 and a β = 0.20, with the estimates of proportion being 0.40 for placebo (P0) and 0.15 for LLLT (P1) a total of 94 patients were evaluated. One-sided test error was the basis for the sample size determination and all the reported P-values were derived from two-sided statistical tests. P-values less than or equal to 0.05 were considered statistically significant; Test type: Superiority or Other; p = 0.05, Chi-squared; Risk Ratio (RR) = 0.158, 95% CI 2-sided [0.050 to 0.498]

2. Secondary Outcome: Oral Mucositis Survival Free, Pain, Opioid Treatment, Hospitalization, Treatment Interruption, Treatment Delay, Patient Weight Loss, Nasogastric Tube or of a Gastrostomy.
Description: Oral mucositis survival free, pain, opioid treatment, hospitalization, treatment interruption, treatment delay, patient weight loss, nasogastric tube or of a gastrostomy.The oral cavities of all patients were evaluated, from the first day to the last day of treatment.
Time Frame: 7 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Placebo | Low Level Laser Therapy
Serious Adverse Events (participants affected / at risk) | 17/47 | 15/47
Other Adverse Events (participants affected / at risk) | 17/47 | 10/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | Low Level Laser Therapy (N=47)
Radiodermatitis (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7) — Unplanned radiotherapy interruptions due to radiodermatis: Laser group = 7 patients and Placebo group = 4 patients
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) — Unplanned radiotherapy interruptions due to pneumonia
Renal and urinary disorders (Renal and urinary disorders) | 5 (5) | 3 (3) — Unplanned chemotherapy interruptions or modification
Ear and labyrinth disorders (Ear and labyrinth disorders) | 3 (3) | 4 (4) — Unplanned chemotherapy interruptions or modification
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 4 (4) | 0 (0) — Unplanned chemotherapy interruptions or modification
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | Low Level Laser Therapy (N=47)
Gastrointestinal disorders (Gastrointestinal disorders) | 17 (17) | 10 (10) — Distribution of severe oral pain intensity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes